CLINICAL TRIAL: NCT05251649
Title: Transcranial Alternating Current Stimulation Combined With 40Hz Sound Stimulation for Treatment of Mild to Moderate Alzheimer's Disease
Brief Title: Transcranial Alternating Current Stimulation Combined With 40Hz Sound Stimulation for Treatment Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhiqi Mao, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChinaPLAGH_LY
Record Dates: First submitted 2022-01-19; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tACS combined with 40 Hz sound stimulation group (Experimental): 15 daily (Monday-Friday) 20min sessions of tACS combined with 40 Hz sound stimulation
  Interventions: Device: tACS combined with 40 Hz sound stimulation
- tACS group (Experimental): 15 daily (Monday-Friday) 20min sessions of tACS stimulation
  Interventions: Device: Transcranial alternating current stimulation
- 40 Hz sound stimulation group (Experimental): 15 daily (Monday-Friday) 20min sessions of 40 Hz sound stimulation
  Interventions: Device: 40 Hz sound stimulation

INTERVENTIONS:
Device: tACS combined with 40 Hz sound stimulation — The tACS instrument (model: XPNS208-B). Two electrodes are placed in the dorsolateral prefrontal cortex and the contralateral supraorbital area. and connected to the tACS device via a thin cable. The intervention will be performed using tACS (40 Hz, 1.5 mA) for 15 sessions of 20 min over 3 weeks (21 days).
  Sound stimulation apparatus: Two sponge earplugs were placed in the ears and the sound stimulator was set to (40Hz, 60dB). Sound stimulation was turned on simultaneously at the beginning of tACS. The duration of sound stimulation was set to 5 min stimulation, 5 min rest, 5 min stimulation, 1 min rest, and continued stimulation until the end of electrical stimulation while sound stimulation was turned off.
  Arms: tACS combined with 40 Hz sound stimulation group
Device: Transcranial alternating current stimulation — The tACS instrument (model: XPNS208-B). Two electrodes are placed in the dorsolateral prefrontal cortex and the contralateral supraorbital area. and connected to the tACS device via a thin cable. The intervention will be performed using tACS (40 Hz, 1.5 mA) for 15 sessions of 20 min over 3 weeks (21 days).
  Arms: tACS group
Device: 40 Hz sound stimulation — Sound stimulation apparatus: Two sponge earplugs were placed in the ears and the sound stimulator was set to (40Hz, 60dB). The duration of the sound stimulation was set to stimulate for 5 min, rest for 5 min, stimulate for 5 min, rest for 1 min, and last for a total of 20 min. 15 sessions of 20 min were performed over a period of 3 weeks (21 days).
  Arms: 40 Hz sound stimulation group

SUMMARY:
Alzheimer's disease is characterized by progressive cognitive decline, and cognition is associated with cerebral concussion. Previous studies have found reduced gamma energy in the brain of AD patients. Therefore, modulation of gamma activity in AD patients may help improve cognitive function.

The purpose of this study was to investigate the safety and tolerability of transcranial alternating current stimulation (tACS) combined with 40Hz sound stimulation in patients with mild to moderate Alzheimer's disease (AD); to compare the effects of tACS combined with sound stimulation, tACS, and 40Hz sound stimulation on cognition in AD patients; and the effects of tACS combined with sound stimulation, tACS, and 40Hz sound stimulation on brain network connectivity in AD patients before and after tACS.

DETAILED DESCRIPTION:
The number of people with Alzheimer's disease is increasing every year, but the available drugs are not effective. Both transcranial alternating current stimulation (tACS) and sound stimulation are non-invasive methods to modulate Central Nervous System excitability. tACS has been shown to modulate cognitive processes by affecting intrinsic oscillatory manipulation and entrainment in the brain. And 40 Hz sound stimulation reduces Aβ amyloid deposition in the hippocampus of AD mice.

Sixty patients with mild-to-moderate AD will be recruited in this randomized, double-blind, controlled study. The researchers will evaluate whether tACS (40Hz) to the DLPFC region or 40Hz sound stimulation to both ears improves cognition in patients with mild to moderate AD. The study will also investigate which stimulation method has a more pronounced and sustained improvement in cognition in the following three groups of patients.

Subjects will be randomized into three groups, with the first group receiving tACS combined with sound stimulation, the second group receiving tACS alone, and the third group receiving sound stimulation alone. All will receive three weeks (15 sessions) of treatment. Patients will be assessed by neuropsychological testing at baseline, post-treatment (21 days) and at the 3-month follow-up. Subjects will be compared by functional MRI at baseline and post-treatment for brain network connectivity before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years, male or female;
2. Meet the diagnosis AD formulated by the National Institute on Aging and the Alzheimer's Association (NIA-AA) dementia diagnostic criteria;
3. Clinical Dementia Rating Scale (CDR) =1.0 or 2.0;
4. MMSE score ≤ 24;
5. Able to move freely or with the aid of a walker or crutches;
6. Good vision and hearing, able to cooperate with examination and treatment;
7. Subjects voluntarily joined and had a guardian to sign the informed consent.

Exclusion Criteria:

1. The presence of preoperative structural brain abnormalities (such as tumors, cerebral infarction, hydrocephalus or intracranial hemorrhage);
2. The presence of other neurological disorders such as multiple sclerosis, epilepsy, Parkinson's disease, etc;
3. Psychiatric system disorders: such as anxiety disorders, affective disorders such as depression, or pharmacogenic psychiatric disorders;
4. Severe medical illness, current use of respiratory medications, cardiovascular medications, anticonvulsants or psychoactive drugs and clinically significant gastrointestinal, renal, hepatic, respiratory, infectious, endocrine or cardiovascular disease, cancer, alcoholism or drug addiction;
5. Severe hearing and visual impairment;
6. Patients with clinical comorbidities with a life expectancy of less than 2 years;
7. Patients who have undergone cranial surgery;
8. Contraindications to undergoing magnetic resonance imaging or receiving transcranial alternating current stimulation (pacemakers, post DBS surgery);
9. Eczema or sensitive skin;
10. Familial Alzheimer's disease;
11. Presence of other types of dementia: vascular dementia, Lewy body dementia, frontotemporal dementia, infectious dementia, etc;
12. Other conditions that, in the opinion of the investigator, may not be suitable for this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale cognitive subscale scores | up to 21 days (end of intervention) ,3 months
  ADAS-cog 11 scale ranges from 0 to 70, and higher value represents a worse outcome. This study will use ADAS-cog to assess changes in the global cognitive function after intervention.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment scores | up to 21 days (end of intervention) ,3 months
  Montreal Cognitive Assessment (MoCA) will be used to evaluate the general cognitive function. MoCA ranges from 0 to 30, and higher value represents a better outcome.
Change in Mini-mental State Examination scores | up to 21 days (end of intervention) ,3 months
  Mini-mental State Examination (MMSE) will be used to evaluate the general cognitive function. MMSE ranges from 0 to 30, and higher value represents a better outcome.
Change in Clinical Dementia Rating scores | up to 21 days (end of intervention) ,3 months
  Clinical Dementia Rating(CDR) will be used to evaluate the level of dementia in AD patients. Mild dementia CDR: 1.0; Moderate dementia CDR: 2.0; Severe dementia CDR: 3.0.
Change in Auditory Verbal Learning Test scores | up to 21 days (end of intervention) ,3 months
  auditory verbal learning test（AVLT）will be used to evaluate the memory function. AVLT ranges from 0 to 36, and higher values representing better outcome.
Change in Boston Naming Test scores | up to 21 days (end of intervention), 3 months
  Boston Naming Test（BNT-30） will be used to assess language function. It ranges from 0 to 30, and higher value represents a better outcome.
Change in Neuropsychiatric Inventory (NPI) scores | up to 21 days (end of intervention), 3 months
  The Neuropsychiatric Inventory will be used to measure neuropsychiatric symptoms. It ranges from 0 to 144, and higher value represents a worse outcome.
Change in Activities of Daily Living scores | up to 21 days (end of intervention), 3 months
  Activities of Daily Living (ADL) scale will be used to assess the change of life quality. It ranges from 20 to 80. The "20" represents normal life ability and the higher score presents the worse life ability.
Change in Magnetic Resonance Imaging performance | up to 21 days (end of intervention), 3 months
  Function Magnetic Resonance Imaging (fMRI) will be used to measure changes in brain connectivity；Structural Magnetic Resonance Imaging (sMRI) will be used to measures structural changes in the brain.
Incidence of tACS Adverse events | up to 21 days (end of intervention), 3 months
  Adverse Events as a result of tACS stimulation will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqi Mao, Ph.D, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

REFERENCES:
- [Derived] Liu Y, Liu S, Tang C, Tang K, Liu D, Chen M, Mao Z, Xia X. Transcranial alternating current stimulation combined with sound stimulation improves cognitive function in patients with Alzheimer's disease: Study protocol for a randomized controlled trial. Front Aging Neurosci. 2023 Jan 9;14:1068175. doi: 10.3389/fnagi.2022.1068175. eCollection 2022. PMID 36698862
- [Derived] Liu Y, Tang C, Wei K, Liu D, Tang K, Chen M, Xia X, Mao Z. Transcranial alternating current stimulation combined with sound stimulation improves the cognitive function of patients with Alzheimer's disease: A case report and literature review. Front Neurol. 2022 Sep 23;13:962684. doi: 10.3389/fneur.2022.962684. eCollection 2022. PMID 36212652